CLINICAL TRIAL: NCT03753997
Title: A Randomized Trial of Diabetes-educated Psychologist to Improve HbA1c and Reduce Diabetes-related Distress
Brief Title: A Trial of Diabetes-educated Psychologist to Improve HbA1c and Reduce Diabetes-related Distress
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Psychologystudy
Record Dates: First submitted 2018-11-21; First posted 2018-11-27 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Type1diabetes; Psychology Functional Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional therapy (No Intervention): Patiens´s will come to the clinic for regular contact with a diabetes nurse.
- Treatment by a Psychologist (Experimental): Patients will meet with a diabetes educated psychologist over 9 months and will come to the clinic for regular contact with a diabetes nurse
  Interventions: Behavioral: Treatment by a diabetes educated psychologist

INTERVENTIONS:
Behavioral: Treatment by a diabetes educated psychologist — Patients will meet a diabetes educated psychologist. There will be a minimum of 5 meetings during the first 3 months and then in the following 6 months there will be a minimum of 2 meetings. More meetings will be scheduled if needed.
  Arms: Treatment by a Psychologist

SUMMARY:
Type 1 diabetes is associated with a significant increase in mortality, cardiovascular disease, injuries on eyes and kidneys. These risks are largely dependent on glycemic control. Multiple strategies of achieving good glycemic control exist. Despite this, only about 20 % of patients in Sweden reach the target HbA1c of ≤ 52 mmol/mol.

It is well-known that when the motivation is high, a large proportion of patients reach good glycaemic control with current treatments, e.g. most pregnant women reach a much better glycaemic control. The patient is then motivated to a greater extent in managing the disease, e.g. by carefully dosing insulin and more closely monitoring blood glucose levels.

Moreover, besides lack of motivation, specific psychiatric conditions are well-known barriers in being compliant with treatments such as depression, eating disorders and attention deficit disorders (ADHD). Further, identified specific diabetes-related psychosocial factors include severe fear of hypoglycaemia, diabetes-burnout, unrealistic treatment goals, poor relationship with physician, feelings of powerlessness and treatment skepticism. These parameters can be measured via a diabetes distress scale where a high score is correlated to higher HbA1c.

The majority of outpatient diabetes clinics in Sweden today request the resource of a diabetes-educated psychologist. However, more evidence is needed from randomized multicentre trials whether such a resource would help to improve HbA1c, reduce diabetes-related distress and improve quality of life.

The primary aim of the current study is to evaluate whether the assistance of a diabetes-educated psychologist in the diabetes care of patients with type 1 diabetes improves HbA1c. Secondary endpoints include studying its influence on diabetes-related distress and quality of life. The study is a 1 year randomized trial where the intervention group will meet with a diabetes-educated psychologist in addition to conventional care.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before trial-related activities (i.e., any activity that would not have been performed during routine patient management)
* Clinical diagnosis of Type 1 diabetes
* Adult patients over 18 years of age
* HbA1c > 62 mmol/mol

Exclusion Criteria:

* Type 2 diabetes
* Diabetes duration <1 year
* Long-term Systemic glucocorticoid treatment during the last 3 months
* Changed treatment the last 3 months regarding MDI vs. Insulin pump or added or stopped CGM or FGM therapy
* Current or planned pregnancy or breastfeeding during the next 12 months
* Planned move during the next 12 months making it not possible to participate in study activities
* Other reason determined by the investigator not being appropriate for participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c from baseline to 52 weeks follow-up | 52 weeks

SECONDARY OUTCOMES:
Change in Diabetes distress scale score from baseline to week 52 | 52 weeks
  Diabetes Distress scale is a questionnaire with 28 questions where patients answer on a scale between 1-6.
Change in quality of life score (ADDQoL) from baseline to week 52 | 52 weeks
  ADDQoL (actual name for questionnaire) is a quality of life questionnaire with 19 questions. Answers are on a scale of 1-4,1-5,1-6 and 1-7
score of Diabetes Treatment satisfaction questionnaire - change (DTSQc) at week 52 | 52 weeks
  8 questions which patients answer on a scale of -3 to 3

OTHER OUTCOMES:
Change in the Diabetes Treatment satisfaction questionnaire - status (DTSQs) score from baseline to week 52 | 52 weeks
  8 questions which patients answer on a scale of 6 to 0
Change in the score of the hypoglycaemia confidence questionnaire from baseline to week 52 | 52 weeks
  9 questions with 4 answer possibilities. Not confident at all, to very confident
Proportion of patients with HbA1c less than 59 mmol/mol at week 52 | 52 weeks
Proportion of patients with HbA1c less than 53 mmol/mol at week 52 | 52 weeks
Proportion of patients lowering HbA1c 5 mmol/mol or more from baseline to week 52 | 52 weeks
Change in total insulin dose from baseline to week 52 | 52 weeks
change weight from baseline to week 52 | 52 weeks
Change in systolic and diastolic blood pressure from baseline to week 52 | 52 week
  Change in systolic and diastolic blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Lind, PhD, Principal Investigator — NU-Hospital Organization, Sweden
Locations (1):
- NU Hospital Group, Uddevalla, Sweden

REFERENCES:
- [Derived] Zeijlemaker J, Anderbro T, Sterner Isaksson S, Lind M. Design and methods of a multicenter randomized clinical trial of effects of diabetes-educated psychologist on glucose management and diabetes distress. Front Clin Diabetes Healthc. 2025 Apr 16;6:1549234. doi: 10.3389/fcdhc.2025.1549234. eCollection 2025. PMID 40308292